CLINICAL TRIAL: NCT03691415
Title: Evaluation of the Safety and Effectiveness of BELKYRA® Inj. for the Treatment of Patients With Submental Fullness Due to Submental Fat: A Post Marketing Surveillance Study in Korea
Brief Title: Evaluation of the Safety and Effectiveness of BELKYRA® Inj. for the Treatment of Patients With Submental Fullness Due to Submental Fat: A Postmarketing Surveillance Study in Korea
Status: Terminated | Type: Observational
Why Stopped: Study discontinued due to business decisions.
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Other Study IDs: CMO-EPI-FAS-0537; EUPAS23762 (Other: EU PAS)
Record Dates: First submitted 2018-09-28; First posted 2018-10-01 (Actual); Last update posted 2020-12-07 (Actual); Status verified 2020-10

CONDITIONS: Submental Fullness
Keywords: Double Chin Fat Reduction
MeSH Terms: interventions — Deoxycholic Acid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- BELKYRA Inj.: Each patient will be administered BELKYRA Inj. at least once and the interval between treatments not less than 1 month apart and follow-up within 3 months of the last treatment session.
  Interventions: Drug: BELKYRA Inj.

INTERVENTIONS:
Drug: BELKYRA Inj. — Patient will be administered BELKYRA Inj. at least once and the interval between treatments not less than 1 month apart.
  Other Names: Deoxycholic acid

SUMMARY:
The purpose of this PMS study is to evaluate the safety and effectiveness of BELKYRA Inj. used according to the dose specified in the instructions for use, for the treatment of patients with SM fullness due to SMF, through active investigation under routine clinical practice

ELIGIBILITY:
Inclusion Criteria:

* Eligible and consenting Korean patients
* Patients who have consented to the study and who have signed the private information protection act form or ICF

Exclusion Criteria:

* Patients having infection at the infection sites
* Patients presenting evidence of causes of enlarged submental area other than localized submental fat (E.g.: thyroid enlargement, enlarged submental salivary glands, cervical lymphadenopathy, etc.)
* Patients participating in an interventional clinical study, currently or within 30 days before enrollment, will not be eligible for inclusion in the study
* Pregnant women
* Renal impairment patients
* Hepatic impairment patients
* Patients with severe laxity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will include adult patient is an adult (≥ 18 years of age) in South Korea treated with BELKYRA for the improvement of moderate to severe convexity or fullness associated with submental fat in adults
Sampling Method: Non-Probability Sample
Enrollment: 71 (Actual)
Dates: Start 2018-09-07 (Actual); Primary Completion 2020-04-14 (Actual); Study Completion 2020-04-14 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Clinician-Reported Submental Fat Rating Scale (CR-SMFRS) | Baseline, Follow up visit (within 3 months of injection)
  A validated scale used by investigators to assess SM convexity/amount of SMF. Specifically, the CR-SMFRS ranges in whole number increments from 0 (absent submental convexity) to 4 (extreme submental convexity)
Change from baseline in Patient-Reported Submental Fat Rating Scale (PR-SMFRS) | Baseline, Follow up visit (within 3 months of injection)
  Validated scale used by patients to evaluate SM size. Specifically, the PR-SMFRS asks patients to assess how much fat they have under their chins by selecting options ranging from "no chin fat at all" to "a very large amount of chin fat".

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne St. Rose, DVM, MSc, PhD, Study Director — Allergan
Locations (4):
- South Korea (4):
  - Oracle-Dermatology, Daejeon
  - Goldenview plastic surgery, Seoul
  - (Apgujeong) Oracle-Dermatology, Seoul
  - Dream-Dermatology, Seoul

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Additional information on study locations near you may be found at AllerganClinicalTrials.com. For any study not on AllerganClinicalTrials.com, please contact IR-CTRegistration@Allergan.com for assistance." — http://www.allerganclinicaltrials.com/